CLINICAL TRIAL: NCT01626898
Title: HIV Prevention Among Latino MSM: Evaluation of a Locally Developed Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: U01PS001570 (NIH)
Record Dates: First submitted 2012-06-21; First posted 2012-06-25 (Estimated); Last update posted 2016-02-03 (Estimated); Status verified 2016-02

CONDITIONS: Risk Reduction Behavior
MeSH Terms: conditions — Risk Reduction Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- HOLA en Grupos (Experimental): The Spanish language HOLA en Grupos intervention consists of four 4-hour group sessions that combine presentations by facilitators who are trained Latino MSM community members, activities, and scenes from a DVD, and is delivered over a period of two weeks to groups of about 10 participants.
  Interventions: Behavioral: HOLA en Grupos
- General health intervention (Active Comparator): The Spanish language comparison condition consists of four 4-hour group sessions designed to increase participants' knowledge about cancer, diabetes, alcohol abuse, and cardiovascular disease, and is delivered over a period of two weeks to groups of about 10 participants.
  Interventions: Behavioral: General Health intervention (comparison intervention )

INTERVENTIONS:
Behavioral: HOLA en Grupos — HOLA en Grupos consists of four 4-hour group sessions that combine presentations by facilitators who are trained Latino MSM community members, activities, and scenes from a DVD, and is delivered over a period of two weeks to groups of about 10 participants. HOLA en Grupos is designed to increase HIV prevention knowledge, condom use and mastery, decrease barriers to risk reduction (e.g., health-compromising aspects of machismo), enhance sexual negotiation skills, and increase use of HIV testing, counseling, and treatment services among intervention participants.
  Arms: HOLA en Grupos
Behavioral: General Health intervention (comparison intervention ) — The Spanish comparison condition consists of four Spanish-language 4-hour group sessions designed to increase participants' knowledge about cancer, diabetes, alcohol abuse, and cardiovascular disease, and is delivered over a period of two weeks to groups of about 10 participants.
  Arms: General health intervention

SUMMARY:
Wake Forest University is partnering with Chatham Social Health Council (a community-based organization) to conduct a randomized controlled trial to evaluate the efficacy of Hombres Ofreciendo Liderazgo y Apoyo (HOLA) en Grupos (Men Giving Leadership and Support in Groups), a Spanish-language HIV risk behavior intervention for Latino men who have sex with men (MSM) in rural North Carolina.

Participants in the HOLA intervention, when compared to those in the comparison intervention, will report: increased consistent use of condoms during sexual intercourse; increased use of HIV and sexually transmitted disease (STD) counseling, testing, and treatment services; greater knowledge concerning the impact of HIV on communities (including Latino and MSM)and HIV risk behaviors and prevention strategies; more positive attitudes towards abstinence and condom use; increased self-efficacy to use and assert the use of condoms with sex partners; increased condom-use mastery scores; decreased barriers to risk reduction (e.g. health-compromising aspects of machismo); and enhanced partner and provider communication and sexual negotiation skills.

DETAILED DESCRIPTION:
Wake Forest University is partnering with Chatham Social Health Council to conduct a randomized controlled trial to evaluate the efficacy of Hombres Ofreciendo Liderazgo y Apoyo (HOLA) en Grupos (Men Giving Leadership and Support in Groups) HIV risk behavior intervention for Latino men who have sex with men (MSM), ages 18 and over, in rural North Carolina.

The Spanish language HOLA en Grupos was developed by the Chatham Social Health Council in close collaboration and partnership with the local Latino community, including Latino MSM, and representatives from a local community-based participatory research (CBPR) partnership that has been in existence for nearly ten years, and has been delivered by the Council to Latino MSM in an area the includes 6 largely rural counties for two years.

HOLA en Grupos consists of four 4-hour group sessions that combine presentations by facilitators who are trained Latino MSM community members, activities, and scenes from a DVD, and is delivered over a period of two weeks to groups of about 10 participants. HOLA en Grupos was designed to increase HIV prevention knowledge, condom use and mastery, decrease barriers to risk reduction (e.g., health-compromising aspects of machismo), enhance sexual negotiation skills, and increase use of HIV testing, counseling, and treatment services among intervention participants.

The Spanish language comparison condition consists of four 4-hour group sessions designed to increase participants' knowledge about cancer, diabetes, alcohol abuse, and cardiovascular disease, and is delivered over a period of two weeks to groups of about 10 participants. The content focus of the comparison condition reflects the desire of community partners to provide this type of information to community members.

A total of 300 Latino MSM (150 per condition) will be screened and if eligible, recruited in waves of 20 men (10 per condition). Eligible individuals must self-identify as Latino or Hispanic, be ≥ 18 years of age, report MSM behavior since age ≥ 18, and provide informed consent. Individuals who have participated in the HOLA en Grupos, or interventions for Latino heterosexual men (HoMBReS or HoMBReS-2), will be excluded from the study. Study assessments will be conducted at baseline and 6-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Male gender
* Self-identify as Latino or Hispanic
* 18 years of age or older
* Speak Spanish
* Have had sex with another man since attaining age 18
* Have not participated in HOLA, HOLA en Grupos, HoMBReS or other Latino Partnership interventions developed and delivered by the Chatham Social Health Council or Wake Forest University during the past 12 months

Exclusion Criteria:

* Have had sex with at least one woman since attaining age 18 but who have not had sex with at least one man since attaining age 18

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 304 (Actual)
Dates: Start 2012-08; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Increased self-reported consistent use of condoms during sexual intercourse | 6 months post-intervention

SECONDARY OUTCOMES:
Increased self-reported use of HIV and sexually transmitted disease (STD) counseling, testing, and treatment services | 6 months post-intervention

CONTACTS AND LOCATIONS:
Overall Officials: Scott D Rhodes, PhD, Study Director — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

REFERENCES:
- [Derived] Rhodes SD, Alonzo J, Mann L, Song EY, Tanner AE, Arellano JE, Rodriguez-Celedon R, Garcia M, Freeman A, Reboussin BA, Painter TM. Small-Group Randomized Controlled Trial to Increase Condom Use and HIV Testing Among Hispanic/Latino Gay, Bisexual, and Other Men Who Have Sex With Men. Am J Public Health. 2017 Jun;107(6):969-976. doi: 10.2105/AJPH.2017.303814. Epub 2017 Apr 20. PMID 28426301